CLINICAL TRIAL: NCT02800109
Title: Impact of Malaria Infection in Pregnancy on Fetal and Newborn Growth - Child Follow-up Until 2 Years of Age, in Relation to the Fetal Growth
Brief Title: Child Follow-up Until 2 Years
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1504
Record Dates: First submitted 2016-05-27; First posted 2016-06-15 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Malaria; Pregnancy
Keywords: Fetal growth; Newborn growth
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples will consist of a 50 uL of finger prick blood sample at month 3,6,9,12,18 and 24, and a stool sample.
  A buccal swab will be collected at 1 and 2 years.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure the impact of maternal malaria on child growth in the two first years of life in relation to fetal growth.

This study is following a birth cohort of children born to pregnant women enrolled in the study "Impact of malaria infection in pregnancy on fetal and newborn growth" (protocol OXTREC 14 08 and Mahidol 2009-003-01). In this cohort growth monitoring is conducted until 2 years of age using routine anthropometric measurements such as weight, length, arm and head circumference. A few additional tests will enhance the sensitivity of the study outcomes with minimal risk. These tests will include anthropometry, screening, nutrition questionnaire and neurodevelopmental assessment.

This study was funded by Wellcome Trust core funding, grant ref. number Wellcome Trust Major Overseas Program Grant no. 220211 (2020-2025)

DETAILED DESCRIPTION:
This is an existing on-going prospective birth cohort of children born to the pregnant women who had fetal growth assessed during pregnancy. In this cohort an expected 10% of pregnant women will be exposed to malaria while the remaining will be free of malaria. Their offspring are already followed up for growth monitoring from birth until 2 years of age with anthropometric measurements including weight, length, arm and head circumference at each scheduled visit. The investigator would like to enhance the sensitivity of the study outcomes with minimal risk for the child by proposing the following anthropometric and screening tests, nutrition questionnaire, and neurodevelopment assessment. In addition a prospective cohort of children born after study approval will be followed on both protocols. The additional measure include:

* Body fat composition (at birth, and monthly up to 4 months unless weight ≥ 8kg)
* Triceps and subscapular skinfold (at 1 and 2 years)
* Anemia, malaria and soil-transmitted helminths screening (every 3 months in first 12 months and 6-monthly 1-2 years)
* Buccal swab (at 1 and 2 years)
* Neurodevelopment (every 6 months)
* Food questionnaire (at 1 and 2 years)

Summary of results:

The beginning of the recruitment was delayed until the finalization and approval of the translated PIS/ICF; from then on, the recruitment was smooth. Overall, 201 children from the ongoing existing birth cohort were still present and eligible to participate in this part of the study; 173 completed 2 years of FUP 28 were lost. Data and samples from these 173 children were included in the analysis of a large, multi-center, study, the INTERBIO-21st.

The pooled findings show 1. Cognitive development, language, and visual skills at 2 years of age vary according to the trajectories of fetal cranial growth 2. There is a critical window period at 20-25 weeks gestational age when fetal cranial trajectories may diverge and when fetal abdominal circumference growth may accelerate or decelerate 3. Preterm newborn's growth and neurocognitive development vary according to their birth phenotype characteristics (i.e. those classified in the "birth infections" phenotype were at higher risk for poor scoring in fine and gross motor development compared to term newborns) 4. An indication of a greater increase in weight in proportion to height during the 2 first years of life if there was a faltering growth phenotype observed during gestation.

Maternal malaria and anemia's role in the development of children were evaluated specifically for this study site and included all the children followed up to one year of age. Preliminary results show that 48% of children are stunted at 2 years of age and that malaria and anemia independently are significant contributors to the decline in growth z-scores during infancy (manuscript in preparation); that 66% of children have anemia (HCT<33%) in the first year of life, the median age for a first HCT<33% is 4 months of age and that moderate, but not mild anemia in infancy reduces the median neurodevelopment score at year of age. Maternal anemia but not malaria is a factor contributing to increased risk of anemia in infants. Results were presented at local and regional and international conferences and were part of a MSc thesis.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent or legal guardian is willing and able to give informed consent for participation in the study
* Able (in the Investigators opinion) to comply with study requirements

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Medical or congenital complications which would (in the investigator's opinion) make it difficult to comply with study requirements
* Aged older than 2 years

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants in a current birth cohort. For those pregnant women who have not yet delivered (circa n=25), permission for their unborn child to commence participation after delivery will be conducted after ethical approval has been received. For those children who have already been born in the existing birth cohort and less than 2 years of age an invitation to participate will be proposed to the parent or legal guardian after ethical approval has been granted.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The proportion of children with sub-optimal growth by 2 years of age among children born to mother exposed to malaria and those born to mother non-exposed to malaria | up to 2 years of age

SECONDARY OUTCOMES:
The median neurocognitive scores by growth groups and malaria-exposed groups | up to 2 years of age
The median age of onset of anemia by growth groups and malaria-exposed Groups | up to 2 years of age
Characterize of molecular signatures (methylation profile of the DNA) by growth groups and malaria-exposed groups | up to 2 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes